CLINICAL TRIAL: NCT02281071
Title: Microsurgical Instruments and Magnification May Enhance Treatment Outcomes Of Laterally Moved, Coronally Advanced Flap in Miller Class III Isolated Recession Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Onur Ozcelik, Professor doctor PhD, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CukurovaU2
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Gingival Recession, Mucogingival Surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- laterally moved coronally advanced flap microsurgical (Experimental): For the test group (LMCAF-M), the surgical procedures were performed with the aid of a galilean loupe, under 2.5x magnification vision, microsurgical instruments and microsurgical suture material .
  Interventions: Procedure: laterally moved coronally advanced flap with microsurgical instruments and x2.5 loupe
- laterally moved coronally advanced flap macrosurgical (Active Comparator): For the control group (LMCAF), LMCAF was performed with conventional instruments (detaylı) and materials (stur). Loupe magnification, microsurgical instruments and suture material were not used in the control group.
  Interventions: Procedure: laterally moved coronally advanced flap with microsurgical instruments and x2.5 loupe

INTERVENTIONS:
Procedure: laterally moved coronally advanced flap with microsurgical instruments and x2.5 loupe — The recipient area for the laterally moved flap was prepared. When the flap was moved in the distal-mesial direction another short horizontal incision was performed at the most apical extension of this vertical incision. Once the mucogingival line was reached, flap elevation was continued split-thickness. Flap elevation was terminated when it was possible to passively move the flap laterally above the exposed root. Flap was sutured.

SUMMARY:
The benefits of microsurgical approaches in periodontal therapy have been described. The main focus of this study is to determine if using microsurgical LMCAF technique would improve the outcomes of the therapy for the Miller Class III isolated recession-type defects.

Six months results of this study showed that LMCAF with microsurgical approach offered better complete and mean root coverage results over macrosurgical LMCAF technique. The superior effect of microsurgical approach on post-operative morbidity can make this technique more preferable for the patients who expected comfortable postoperative period.

This study supports that using the microsurgical aproach with LMCAF procedure significantly affects the clinical and patient-centered success of treating Miller Class III isolated typed defects.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Miller Class III isolated gingival recessions located at upper and lower incisors and canines (Miller 1985)
* Presence of identifiable cementoenamel junction (CEJ)
* Presence of a step ≤ 2mm at CEJ level and/or the presence of a root abrasion, but with an identifiable CEJ
* Lateral keratinized tissue width at least 6 mm greater than the width of the recession measured at the level of the cemento-enamel junction (CEJ)
* Lateral keratinized tissue height at least 2 mm greater than the buccal probing depth of the adjacent tooth/teeth
* Full-mouth plaque score and full-mouth bleeding score of < 15% (four sites/tooth) -No occlusal interferences; all patients were nonsmokers

Exclusion Criteria:

* Tooth with a prosthetic crown or restoration involving CEJ
* Patients with a history of destructive periodontal disease (o zaman class 3 nasıl oluştu demiş adam) or repeated abscess formation
* Presence of systemic disease or taking medications known to interfere with periodontal tissue health or healing (patients with insulin-dependent diabetes
* History of malignancy, radiotherapy, or chemotherapy for malignancy
* Disease affecting connective tissue metabolism)
* Patient pregnant or nursing during the past 5 months
* Patients who participated in a clinical trial within the past 6 months

Ages: 22 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the percentage of root coverage | at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)